CLINICAL TRIAL: NCT07343310
Title: Multi-Center, Open-label, Single Dosing, Dose-Ascending, Phase 1 Study to Evaluate the Safety and Tolerability of KINE-101 in Patients With CIDP (Chronic Inflammatory Demyelinating Polyneuropathy) Refractory to Corticosteroid Treatment
Brief Title: A First-in-Patient Clinical Trial of KINE-101 in Patients With Corticosteroid-Refractory CIDP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kine Sciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CIDP101-CR1-001P
Record Dates: First submitted 2025-12-10; First posted 2026-01-15 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: CIDP - Chronic Inflammatory Demyelinating Polyneuropathy
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Intervention Model Description: Sequential dose escalation in single experimental arm with cohorts receiving 120 mg, 240 mg, or 360 mg.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- KINE-101 120mg (Experimental): Subjects received a single intravenous dose of KINE-101 120 mg.
  Interventions: Drug: KINE-101
- KINE-101 240 mg (Experimental): Subjects received a single intravenous dose of KINE-101 240 mg.
  Interventions: Drug: KINE-101
- KINE-101 360 mg (Experimental): Subjects received a single intravenous dose of KINE-101 360 mg.
  Interventions: Drug: KINE-101

INTERVENTIONS:
Drug: KINE-101 — KINE-101 injection, 12.5 mg/mL, administered once intravenously on Day 1.

SUMMARY:
This is a multicenter, open-label, single-dose, dose-escalation study evaluating the safety and tolerability of intravenous (IV) KINE-101 in patients with corticosteroid-refractory chronic inflammatory demyelinating polyneuropathy (CIDP). On Day 1, subjects receive a single IV dose of KINE-101 at the assigned cohort level and are discharged on Day 3, approximately 48 hours after investigational product (IP) administration, once all required in-clinic assessments have been completed. Safety assessments (including dose-limiting toxicities [DLTs], adverse events, clinical laboratory tests, vital signs, physical examinations, and 12-lead ECGs), exploratory efficacy evaluations, and PK/PD assessments are conducted through Day 28 in accordance with the schedule of assessments.

Exploratory efficacy assessments through Day 28 include changes from baseline in the following clinical measures: Inflammatory Neuropathy Cause and Treatment (INCAT) disability score, Medical Research Council (MRC) total sum score, Inflammatory Rasch-Built Overall Disability Scale (I-RODS), Timed Up-and-Go (TUG) test, mean grip strength, and the Overall Neuropathy Limitations Scale (ONLS).

Pharmacodynamic (PD) assessments include immunophenotyping of CD4+ T-cell subsets (CD4, CD25, FOXP3, CD39, CD69, CTLA-4, LAG-3, TNFR2, TIGIT, CCR5, and CXCR3); measurement of serum cytokines and immunoglobulins (IgM, IgG, IL-2, IL-6, IL-10, IL-17, IFN-γ, MCP-1, and TGF-β); evaluation of autoantibody and complement markers (antinuclear antibodies, anti-SM, anti-RNP, anti-SSA, anti-double-stranded DNA antibodies, and complement C4); and additional laboratory parameters related to systemic inflammation.

Dose escalation follows a standard 3+3 design based on review of safety, including DLTs, in the preceding cohort. Three KINE-101 dose cohorts are planned: Cohort 1 (120 mg), Cohort 2 (240 mg), and Cohort 3 (360 mg). If safety and tolerability are deemed acceptable in a given cohort, enrollment proceeds sequentially to the next higher dose level.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥19 years at informed consent.
* Diagnosed with CIDP and refractory to corticosteroid treatment for ≥3 months prior to enrollment, or corticosteroid treatment deemed inappropriate or cannot be continued for safety reasons.
* Meets EAN/PNS 2021 criteria for typical CIDP:

  * Progressive or relapsing symmetrical motor weakness in arms and legs with sensory involvement in ≥2 limbs
  * Symptom duration ≥8 weeks
  * Reduced or absent tendon reflexes in all extremities
* INCAT disability score ≥2 at screening (score of 2 must result solely from leg disability).
* CIDP Disease Activity Status (CDAS) score ≥3 at screening.
* Received IVIg ≥2 months prior to IP administration.
* If the subject is of childbearing potential, agrees to use highly effective contraception for ≥28 days after IP administration.
* Adequate venous access for IV administration and blood sampling.
* Willing and able to comply with all study procedures.

Exclusion Criteria:

* Polyneuropathy due to other causes (e.g., MMN, MGUS with anti-MAG antibodies, hereditary neuropathies, POEMS syndrome, diabetic or systemic disease-related neuropathy, drug/toxin-induced neuropathy).
* History of myelopathy or confirmed central demyelination.
* Known allergy or hypersensitivity to the investigational product or its excipients.
* Uncontrolled severe hepatic disease, CNS disorders, alcoholism, substance abuse, or psychiatric disorders.
* Other medical conditions that better explain symptoms (e.g., stroke, CNS trauma, connective tissue disease).
* Malignancy within 5 years, except adequately treated low-risk cancers.
* Moderate to severe heart failure or severe cardiovascular disease (e.g., MI, ischemic stroke).
* Moderate to severe substance or alcohol use disorder within 1 year.
* Positive pregnancy test or planning pregnancy, breastfeeding, or gamete donation within 28 days post-IP.
* Use of systemic immunosuppressants or immunostimulants within 5 half-lives prior to IP administration.
* Plasma exchange within 8 weeks prior to IP administration.
* Chronic infections or expected need for anti-infective treatment during the study.
* Active hepatitis B or C infection or HIV positive.
* Abnormal labs at screening: AST/ALT >3×ULN, Hb <9 g/dL, ANC <1,500/μL, Platelets <100×10³/μL.
* Major surgery within 3 months or planned during study participation.
* Investigator deems subject unsuitable for any reason.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2024-08-27 (Actual); Primary Completion 2025-04-14 (Actual); Study Completion 2025-04-14 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | Day 1 to Day 28
  Incidence, severity, and relationship of treatment-emergent adverse events following a single intravenous dose of KINE-101.
Number of Participants with Clinically Significant Abnormal Hematology | Day 1 to Day 28
  Count of participants with clinically significant abnormal hematology findings (e.g., white blood cell count, hemoglobin, platelets, absolute neutrophil count), as defined per protocol.
Number of Participants with Clinically Significant Abnormal Clinical Chemistry | Day 1 to Day 28
  Count of participants with clinically significant abnormal clinical chemistry findings (e.g., ALT, AST, creatinine), as defined per protocol.
Number of Participants with Clinically Significant Abnormal Urinalysis | Day 1 to Day 28
  Count of participants with clinically significant abnormal urinalysis findings (e.g., protein/albumin, glucose, pH), as defined per protocol.
Number of Participants with Clinically Significant Abnormal Vital Signs | Day 1 to Day 28
  Count of participants with clinically significant abnormal vital sign findings (e.g., systolic or diastolic blood pressure, pulse rate, body temperature, respiratory rate), as defined per protocol.
Number of Participants with Clinically Significant Abnormal Physical Examination | Day 1 to Day 28
  Count of participants with clinically significant abnormal physical examination findings, as defined per protocol.
Number of Participants with Clinically Significant Abnormal Electrocardiogram | Day 1 to Day 28
  Count of participants with clinically significant abnormal electrocardiogram findings (e.g., PR interval, QRS duration, QT interval), as defined per protocol.

OTHER OUTCOMES:
Change From Baseline in Inflammatory Neuropathy Cause and Treatment (INCAT) Disability Score | Day 1 (predose), Day 14, and Day 28
  Change from baseline in the INCAT disability score (range 0-10; higher scores indicate worse disability).
Change From Baseline in Medical Research Council (MRC) Sum Score | Day 1 (predose), Day 14, and Day 28
  Change from baseline in the MRC sum score (range 0-60; higher scores indicate better muscle strength).
Change From Baseline in Inflammatory Rasch-Built Overall Disability Scale (I-RODS) | Day 1 (predose), Day 14, and Day 28
  Change from baseline in the I-RODS score (range 0-48; higher scores indicate better function).
Change From Baseline in Timed Up-and-Go (TUG) Test | Day 1 (predose), Day 14, and Day 28
  Change from baseline in the Timed Up-and-Go test, measured in seconds (lower values indicate better performance).
Change From Baseline in Mean Grip Strength | Day 1 (predose), Day 14, and Day 28
  Change from baseline in mean grip strength (higher values indicate greater muscle strength).
Change From Baseline in Overall Neuropathy Limitations Scale (ONLS) | Day 1 (predose), Day 14, and Day 28
  Change from baseline in the ONLS score (range 0-12; higher scores indicate worse disability).
Peak Plasma Concentration of KINE-101 (Cmax) | Day 1
  Maximum observed plasma concentration of KINE-101.
Area Under the Plasma Concentration-Time Curve of KINE-101 (AUC) | Day 1
  Area under the plasma concentration-time curve of KINE-101 (AUClast and AUCinf).
Change From Baseline in Immunophenotyping markers following KINE-101 administration | Day 1 to Day 28
  The change from baseline in immunophenotyping markers following intravenous administration of KINE-101 including CD4, CD25, FoxP3, CD39, CD69, CTLA4, LAG-3, TNFR2, TIGIT, CCR5, and CXCR3.
Change From Baseline in Serum biomarkers following KINE-101 administration | Day 1 to Day 28
  The change from baseline in serum biomarkers following intravenous administration of KINE-101 including IgG, IgM, IL-2, IL-6, IL-10, IL-17, IFN-gamma, MCP-1, and TGF-beta.
Changes From Baseline in Autoantibodies and Inflammatory Laboratory markers following KINE-101 administration | Day 1 to Day 28
  Changes from baseline in serum autoantibodies and inflammatory laboratory markers.

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Park, Study Director — Kine Sciences Co., Ltd.
Locations (2):
- South Korea (2):
  - Kangbuk Samsung Hospital, Seoul, Seoul
  - Samsung Medical Center, Seoul, Seoul